CLINICAL TRIAL: NCT01793545
Title: Methylation Markers for Natural History and Early Detection of Endometrial Cancer
Brief Title: Endometrial Cancer Testing With Vaginal and Endometrial Cell Samples
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913073; 13-C-N073
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Endometrial Cancer; Gynecological Cancers
Keywords: Endometrial Cancer; Gynecological Cancers; Screening
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Endometrial Cancer Cohort: Women with abnormal bleeding or other conditions associated with increased risk ofendometrial cancer.

SUMMARY:
Background:

- Endometrial cancer is one of the most common gynecologic cancers. If it is caught at an early stage, it can be treated more easily. Women who have this type of cancer often have a history of irregular menstrual bleeding. They may also have abnormal findings during gynecologic exams. Pap smears and cervical cell collection may be able to collect cell samples for cancer testing. However, samples from the vagina or endometrium may produce more accurate results. Researchers want to collect vaginal and endometrial cell samples to improve their tests for and understanding of endometrial cancer.

Objectives:

- To collect vaginal and endometrial cell samples to study endometrial cancer.

Eligibility:

- Women at least 18 years of age who have had symptoms of abnormal uterine or post-menopausal bleeding, or abnormal ultrasound findings.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will have a pelvic exam. Before the exam, they will insert a small tampon in the vagina. The tampon will stay in place for about 10 to 30 minutes. The tampon will then be removed and collected for the study.
* During the pelvic exam, tissue will be collected from the uterine lining with a special brush. An additional sample (biopsy) will be collected from the lining.
* A blood sample will also be collected as part of the study.

DETAILED DESCRIPTION:
Endometrial cancer will account for approximately 47,310 incident cases and 8,010 related deaths in 2012. Most endometrial cancers develop slowly through progression of well characterized precursors, many of which regress with progesterone treatment or are curable with hysterectomy. Thus, early detection of endometrial cancer precursors can prevent many endometrial cancers and reduce mortality. Using DNA methylation profiling in the Polish Endometrial Cancer Study (PECS) and the Benign Reproductive Tissue Evaluation (BRTE) Study, we identified a panel of markers that is strongly and specifically linked to endometrial cancer. Concurrently, we have developed two sampling methods for detecting endometrial cancer and its precursors via DNA methylation analysis: vaginal tampons and endometrial brushings. Preliminary data demonstrate that DNA methylation markers are detectable in tampons and endometrial brushings and can identify women with endometrial cancer. We propose to extend the effort by collecting vaginal tampons and endometrial brushings from about 2000 women who are at increased risk of endometrial cancer and who present at the Mayo Clinic Division of Medical Gynecology. We will test our candidate panel of DNA methylation markers in this population and evaluate the clinical performance to detect endometrial hyperplasia and endometrial cancer. Success of this project could lead to development of early detection tests, including self-sampling strategies that would improve management of abnormal vaginal bleeding, endometrial cancer and its precursors.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women should meet at least one of the following criteria:

* Abnormal uterine bleeding
* Postmenopausal bleeding
* Thickened endometrial stripe
* Hereditary predisposition to endometrial cancer (e.g. HNPCC)
* Women referred for endometrial biopsy to evaluate suspicion or high risk of endometrial cancer

EXCLUSION CRITERIA:

* Prior hysterectomy
* Pregnant women (There will be a verbal screen by the clinic nurse and the physician about a potential pregnancy and a pregnancy test may be conducted if there is any doubt)
* Prior pelvic radiation
* Cervical stenosis that renders Tao brush sampling impossible

Ages: 45 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with abnormal bleeding or other conditions associated with increased risk of endometrial cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1932 (Actual)
Dates: Start 2013-02-11 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Endometrial Cancer and Endometrial Hyper Plasia | 1 to 5 years
  Histologically confirmed endometrial cancer or endometrial hyperplasia

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Wentzensen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Mayo Clinic, Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Armstrong K, Randall TC, Polsky D, Moye E, Silber JH. Racial differences in surgeons and hospitals for endometrial cancer treatment. Med Care. 2011 Feb;49(2):207-14. doi: 10.1097/MLR.0b013e3182019123. PMID 21150796
- [Background] Dimitraki M, Tsikouras P, Bouchlariotou S, Dafopoulos A, Liberis V, Maroulis G, Teichmann AT. Clinical evaluation of women with PMB. Is it always necessary an endometrial biopsy to be performed? A review of the literature. Arch Gynecol Obstet. 2011 Feb;283(2):261-6. doi: 10.1007/s00404-010-1601-3. Epub 2010 Aug 4. PMID 20683604
- [Background] Lacey JV Jr, Ioffe OB, Ronnett BM, Rush BB, Richesson DA, Chatterjee N, Langholz B, Glass AG, Sherman ME. Endometrial carcinoma risk among women diagnosed with endometrial hyperplasia: the 34-year experience in a large health plan. Br J Cancer. 2008 Jan 15;98(1):45-53. doi: 10.1038/sj.bjc.6604102. Epub 2007 Nov 20. PMID 18026193